CLINICAL TRIAL: NCT00991276
Title: A Randomized, Double-Blind, Placebo-Controlled, 3-Way Crossover, Multicenter Polysomnography Study Of Pregabalin And Pramipexole In Adults With Restless Legs Syndrome
Brief Title: Polysomnography Study Of Pregabalin And Pramipexole Versus Placebo In Patients With Restless Legs Syndrome And Associated Sleep Disturbance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081185
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Results first posted 2012-10-08 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2012-09

CONDITIONS: Restless Legs Syndrome
Keywords: restless legs syndrome RLS polysomnography PSG sleep disturbance patient reported outcome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pregabalin; Pramipexole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- pregabalin (Experimental)
  Interventions: Drug: pregabalin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- pramipexole (Active Comparator)
  Interventions: Drug: pramipexole

INTERVENTIONS:
Drug: pregabalin — capsules; 300 mg once-per-day; 4 weeks of treatment
  Other Names: Lyrica
  Arms: pregabalin
Drug: placebo — capsules; 0 mg once-per-day; 4 weeks of treatment
  Arms: placebo
Drug: pramipexole — capsules; 0.5 mg once-per-day; 4 weeks of treatment
  Other Names: Mirapex
  Arms: pramipexole

SUMMARY:
The purpose of this study is to assess the efficacy and safety of pregabalin and pramipexole versus placebo in the treatment of restless legs syndrome and associated sleep disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of restless legs syndrome with a total score of 15 or more points on the International RLS rating scale (IRLS).
* RLS symptoms interfering with sleep on 3 or more nights per week for at least 6 months.
* PSG confirmation of WASO of at least 60 min, PLMI of 10 or more, and total sleep time of at least 3 hrs and less than 6.5 hrs.

Exclusion Criteria:

* Secondary RLS.
* Daytime RLS symptoms requiring treatment.
* Primary sleep disorder.
* Sleep apnea.
* Night or shift work.
* Concurrent medical disorder that could interfere with efficacy assessment or present a safety concern.
* Pregnant or lactating women.
* Women of child-bearing potential not using acceptable method of birth control.
* Use of prohibited medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (38):
  - Pfizer Investigational Site, Jasper, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Burlingame, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Redlands, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Hallandale, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Spring Hill, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Chevy Chase, Maryland
  - Pfizer Investigational Site, Brighton, Massachusetts
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Portage, Michigan
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Dublin, Ohio
  - Pfizer Investigational Site, Middleburg Heights, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Clarks Summit, Pennsylvania
  - Pfizer Investigational Site, Lafayette Hill, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas

REFERENCES:
- [Derived] Garcia-Borreguero D, Patrick J, DuBrava S, Becker PM, Lankford A, Chen C, Miceli J, Knapp L, Allen RP. Pregabalin versus pramipexole: effects on sleep disturbance in restless legs syndrome. Sleep. 2014 Apr 1;37(4):635-43. doi: 10.5665/sleep.3558. PMID 24899755
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081185&StudyName=Polysomnography%20Study%20Of%20Pregabalin%20And%20Pramipexole%20Versus%20Placebo%20In%20Patients%20With%20Restless%20Legs%20Syndrome%20And%20Associated%20Sleep%20Disturbance

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Pramipexole 0.5 mg Then Pregabalin 300 mg: Placebo (PBO) capsule matched to pramipexole (PPX) 0.5 milligram (mg) once daily or pregabalin (PGB) 300 mg once daily (matching placebo escalation and tapering scheme was followed) in first intervention period then PPX capsule 0.5 mg once daily following a 2 week up escalation, Day 1-5: 0.125 mg; Day 6-10: 0.25 mg and Day 11 onwards: 0.5 mg fixed dose for 19 days followed by tapering schedule (Day 1-3: 0.25 mg and Day 4-6: 0.125 mg) in second intervention period and PGB capsule 300 mg once daily following a 2 week up escalation, Day 1-5: 75 mg; Day 6-10: 150 mg and Day 11 onwards: 300 mg fixed dose for 19 days followed by tapering schedule (Day 1-3: 150 mg and Day 4-6: 75 mg) in third intervention period. A PBO wash-out period of 7 days was maintained between each period.
- Pramipexole 0.5 mg Then Pregabalin 300 mg Then Placebo: PPX capsule 0.5 mg once daily following a 2 week up escalation, Day 1-5: 0.125 mg; Day 6-10: 0.25 mg and Day 11 onwards: 0.5 mg fixed dose for 19 days followed by tapering schedule (Day 1-3: 0.25 mg and Day 4-6: 0.125 mg) in first intervention period then PGB capsule 300 mg once daily following a 2 week up escalation, Day 1-5: 75 mg; Day 6-10: 150 mg and Day 11 onwards: 300 mg fixed dose for 19 days followed by tapering schedule (Day 1-3: 150 mg and Day 4-6: 75 mg) in second intervention period and PBO capsule matched to PPX 0.5 mg once daily or PGB 300 mg once daily (matching placebo escalation and tapering scheme was followed) in third intervention period. A PBO wash-out period of 7 days was maintained between each period.
- Pregabalin 300 mg Then Placebo Then Pramipexole 0.5 mg: PGB capsule 300 mg once daily following a 2 week up escalation, Day 1-5: 75 mg; Day 6-10: 150 mg and Day 11 onwards: 300 mg fixed dose for 19 days followed by tapering schedule (Day 1-3: 150 mg and Day 4-6: 75 mg) in first intervention period then PBO capsule matched to PPX 0.5 mg once daily or PGB 300 mg once daily (matching placebo escalation and tapering scheme was followed) in second intervention period and PPX capsule 0.5 mg once daily following a 2 week up escalation, Day 1-5: 0.125 mg; Day 6-10: 0.25 mg and Day 11 onwards: 0.5 mg fixed dose for 19 days followed by tapering schedule (Day 1-3: 0.25 mg and Day 4-6: 0.125 mg) in third intervention period. A PBO wash-out period of 7 days was maintained between each period.
- Pregabalin 300 mg Then Pramipexole 0.5 mg Then Placebo: PGB capsule 300 mg once daily following a 2 week up escalation, Day 1-5: 75 mg; Day 6-10: 150 mg and Day 11 onwards: 300 mg fixed dose for 19 days followed by tapering schedule (Day 1-3: 150 mg and Day 4-6: 75 mg) in first intervention period then PPX capsule 0.5 mg once daily following a 2 week up escalation, Day 1-5: 0.125 mg; Day 6-10: 0.25 mg and Day 11 onwards: 0.5 mg fixed dose for 19 days followed by tapering schedule (Day 1-3: 0.25 mg and Day 4-6: 0.125 mg) in second intervention period and PBO capsule matched to PPX 0.5 mg once daily or PGB 300 mg once daily (matching placebo escalation and tapering scheme was followed) in third intervention period. A PBO wash-out period of 7 days was maintained between each period.
- Placebo Then Pregabalin 300 mg Then Pramipexole 0.5 mg: PBO capsule matched to PPX 0.5 mg once daily or PGB 300 mg once daily (matching placebo escalation and tapering scheme was followed) in first intervention period then PGB capsule 300 mg once daily following a 2 week up escalation, Day 1-5: 75 mg; Day 6-10: 150 mg and Day 11 onwards: 300 mg fixed dose for 19 days followed by tapering schedule (Day 1-3: 150 mg and Day 4-6: 75 mg) in second intervention period and PPX capsule 0.5 mg once daily following a 2 week up escalation, Day 1-5: 0.125 mg; Day 6-10: 0.25 mg and Day 11 onwards: 0.5 mg fixed dose for 19 days followed by tapering schedule (Day 1-3: 0.25 mg and Day 4-6: 0.125 mg) in third intervention period. A PBO wash-out period of 7 days was maintained between each period.
- Pramipexole 0.5 mg Then Placebo Then Pregabalin 300 mg: PPX capsule 0.5 mg once daily following a 2 week up escalation, Day 1-5: 0.125 mg; Day 6-10: 0.25 mg and Day 11 onwards: 0.5 mg fixed dose for 19 days followed by tapering schedule (Day 1-3: 0.25 mg and Day 4-6: 0.125 mg) in first intervention period then PBO capsule matched to PPX 0.5 mg once daily or PGB 300 mg once daily (matching placebo escalation and tapering scheme was followed) in second intervention period and PGB capsule 300 mg once daily following a 2 week up escalation, Day 1-5: 75 mg; Day 6-10: 150 mg and Day 11 onwards: 300 mg fixed dose for 19 days followed by tapering schedule (Day 1-3: 150 mg and Day 4-6: 75 mg) in third intervention period. A PBO wash-out period of 7 days was maintained between each period.
Period: First Intervention Period
Arm/Group | Placebo Then Pramipexole 0.5 mg Then Pregabalin 300 mg | Pramipexole 0.5 mg Then Pregabalin 300 mg Then Placebo | Pregabalin 300 mg Then Placebo Then Pramipexole 0.5 mg | Pregabalin 300 mg Then Pramipexole 0.5 mg Then Placebo | Placebo Then Pregabalin 300 mg Then Pramipexole 0.5 mg | Pramipexole 0.5 mg Then Placebo Then Pregabalin 300 mg
Started | 15 | 13 | 14 | 15 | 15 | 13
Completed | 15 | 10 | 14 | 11 | 11 | 12
Not Completed | 0 | 3 | 0 | 4 | 4 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Insufficient clinical response | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0 | 0
Period: Placebo Wash-out Period (7 Days)
Arm/Group | Placebo Then Pramipexole 0.5 mg Then Pregabalin 300 mg | Pramipexole 0.5 mg Then Pregabalin 300 mg Then Placebo | Pregabalin 300 mg Then Placebo Then Pramipexole 0.5 mg | Pregabalin 300 mg Then Pramipexole 0.5 mg Then Placebo | Placebo Then Pregabalin 300 mg Then Pramipexole 0.5 mg | Pramipexole 0.5 mg Then Placebo Then Pregabalin 300 mg
Started | 15 | 10 | 14 | 11 | 11 | 12
Completed | 15 | 10 | 14 | 11 | 11 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | Placebo Then Pramipexole 0.5 mg Then Pregabalin 300 mg | Pramipexole 0.5 mg Then Pregabalin 300 mg Then Placebo | Pregabalin 300 mg Then Placebo Then Pramipexole 0.5 mg | Pregabalin 300 mg Then Pramipexole 0.5 mg Then Placebo | Placebo Then Pregabalin 300 mg Then Pramipexole 0.5 mg | Pramipexole 0.5 mg Then Placebo Then Pregabalin 300 mg
Started | 15 | 10 | 14 | 11 | 11 | 12
Completed | 14 | 8 | 14 | 9 | 10 | 11
Not Completed | 1 | 2 | 0 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 1
Period: Placebo Wash-out Period (7 Days)
Arm/Group | Placebo Then Pramipexole 0.5 mg Then Pregabalin 300 mg | Pramipexole 0.5 mg Then Pregabalin 300 mg Then Placebo | Pregabalin 300 mg Then Placebo Then Pramipexole 0.5 mg | Pregabalin 300 mg Then Pramipexole 0.5 mg Then Placebo | Placebo Then Pregabalin 300 mg Then Pramipexole 0.5 mg | Pramipexole 0.5 mg Then Placebo Then Pregabalin 300 mg
Started | 14 | 8 | 14 | 9 | 10 | 11
Completed | 14 | 8 | 14 | 9 | 10 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | Placebo Then Pramipexole 0.5 mg Then Pregabalin 300 mg | Pramipexole 0.5 mg Then Pregabalin 300 mg Then Placebo | Pregabalin 300 mg Then Placebo Then Pramipexole 0.5 mg | Pregabalin 300 mg Then Pramipexole 0.5 mg Then Placebo | Placebo Then Pregabalin 300 mg Then Pramipexole 0.5 mg | Pramipexole 0.5 mg Then Placebo Then Pregabalin 300 mg
Started | 14 | 8 | 14 | 9 | 10 | 11
Completed | 13 | 8 | 13 | 8 | 10 | 10
Not Completed | 1 | 0 | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Pramipexole 0.5 mg Then Pregabalin 300 mg | Pramipexole 0.5 mg Then Pregabalin 300 mg Then Placebo | Pregabalin 300 mg Then Placebo Then Pramipexole 0.5 mg | Pregabalin 300 mg Then Pramipexole 0.5 mg Then Placebo | Placebo Then Pregabalin 300 mg Then Pramipexole 0.5 mg | Pramipexole 0.5 mg Then Placebo Then Pregabalin 300 mg | Total
Number analyzed (Participants) | 15 | 13 | 14 | 15 | 15 | 13 | 85
Age, Customized [Number; unit: participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 to 44 years | 3 | 4 | 1 | 2 | 5 | 3 | 18
  45 to 64 years | 8 | 7 | 11 | 10 | 8 | 8 | 52
  Greater than or equal to 65 years | 4 | 2 | 2 | 3 | 2 | 2 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 8 | 9 | 12 | 7 | 54
  Male | 4 | 6 | 6 | 6 | 3 | 6 | 31

OUTCOME MEASURES:

1. Primary Outcome: Wake After Sleep Onset (WASO)
Description: WASO as determined by Polysomnography (PSG) was time spent awake from sleep onset to final awakening. WASO= Wake Time During Sleep [WTDS] epochs + Wake Time After Sleep [WTAS] epochs)/2. WTDS: number of wake epochs (30 seconds of PSG recording) after onset of persistent sleep and prior to final awakening or end of 8-hour recording/2 and WTAS: number of wake epochs after final awakening until end of the 8-hour recording/2. WASO was measured on 2 consecutive days within a period. Arithmetic mean of WASO of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: Week 5 (End of Intervention Period 1), Week 11 (End of Intervention Period 2) and Week 17 (End of Intervention Period 3) or Early Termination (ET)
Population: Intent to Treat (ITT) population included set of randomized participants who had at least 1 dose of study medication and had at least 1 post-randomization efficacy assessment. 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Groups:
- Pregabalin 300 mg: PGB capsule 300 mg once daily in any intervention period.
- Pramipexole 0.5 mg: PPX capsule 0.5 mg once daily in any intervention period.
- Placebo: PBO capsule matched to PPX 0.5 mg once daily or PGB 300 mg once daily in any intervention period.
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
minutes | 51.50 [43.20 to 59.79] | 78.42 [70.34 to 86.51] | 78.60 [70.29 to 86.90]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The least squares (LS) means and standard errors (SE) were used to test for a treatment difference and construct 2-sided 95% confidence intervals (CIs). The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — This analysis was step 1 in a step-down procedure (if p-value < 0.05, then continue to next step) used to control the Type I error rate; LS Mean Difference = -27.10, 95% CI 2-sided [-35.78 to -18.42], Standard Error of Mean 4.38
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — This analysis was not included in the step-down procedure (if p-value < 0.05, then continue to next step) to control Type I error; LS Mean Difference = -26.93, 95% CI 2-sided [-35.54 to -18.32], Standard Error of Mean 4.35
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9684, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.17, 95% CI 2-sided [-8.72 to 8.38], Standard Error of Mean 4.32

2. Secondary Outcome: Periodic Limb Movement Arousal Index (PLMAI)
Description: PLMAI, as determined by PSG was number of periodic limb movements leading to arousal per hour (per hour of Total Sleep Time [TST]). Arithmetic mean of PLMAI of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: Week 5 (End of Intervention Period 1), Week 11 (End of Intervention Period 2) and Week 17 (End of Intervention Period 3) or ET
Population: ITT population included set of randomized participants who had at least 1 dose of study medication and had at least one post-randomization efficacy assessment. 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: movement/hour
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
movement/hour | 3.93 [2.49 to 5.36] | 2.66 [1.27 to 4.06] | 7.61 [6.17 to 9.04]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — This analysis was step 2 in a step-down procedure (if p-value < 0.05, then continue to next step) used to control the Type I error rate; LS Mean Difference = -3.68, 95% CI 2-sided [-5.44 to -1.92], Standard Error of Mean 0.89
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1541, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 1.26, 95% CI 2-sided [-0.48 to 3.01], Standard Error of Mean 0.88
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -4.94, 95% CI 2-sided [-6.68 to -3.21], Standard Error of Mean 0.88

3. Secondary Outcome: Subjective Total Sleep Time (sTST)
Description: sTST as derived from Subjective Sleep Questionnaire (SSQ), a participant reported subjective estimate of the total amount of time the participant was asleep after lights out until final awakening. Completed by the participant 30 minutes after waking; recall period is the night before. Arithmetic mean of sTST of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: Week 3 and Week 5 of Each Intervention Period or ET
Population: ITT population included set of randomized participants who had at least 1 dose of study medication and had at least 1 post-randomization efficacy assessment. 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 72 | 70
minutes | 400.97 [386.36 to 415.58] | 374.19 [360.00 to 388.37] | 370.16 [355.69 to 384.63]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — This analysis was step 3 in a step-down procedure (if p-value < 0.05, then continue to next step) used to control the Type I error rate; LS Mean Difference = 30.81, 95% CI 2-sided [16.14 to 45.49], Standard Error of Mean 7.42
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 26.79, 95% CI 2-sided [12.26 to 41.32], Standard Error of Mean 7.34
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5807, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 4.03, 95% CI 2-sided [-10.36 to 18.41], Standard Error of Mean 7.27

4. Secondary Outcome: Minutes of Stage N1, N2, N3 and R Sleep
Description: Minutes of Stage 1 Non-Rapid Eye Movement (Non-REM) sleep (Stage N1), Stage 2 Non-REM sleep (Stage N2), Stage 3 Non-REM sleep (Stage N3) or Slow Wave Sleep (SWS) and Stage REM (Stage R) sleep, as determined by PSG were calculated as total number of Stage N1 30-second (30-sec) epochs divided by 2, total number of Stage N2 30-sec epochs divided by 2, total number of Stage N3 30-sec epochs divided by 2 and total number of Stage R 30-sec epochs divided by 2 respectively. Arithmetic mean of minutes of stage N1, N2, N3 and R sleep of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
minutes
  Stage N1 Sleep | 38.06 [32.97 to 43.14] | 48.38 [43.38 to 53.38] | 43.72 [38.63 to 48.81]
  Stage N2 Sleep | 227.05 [215.01 to 239.09] | 241.52 [229.76 to 253.27] | 204.35 [192.29 to 216.40]
  Stage N3 Sleep/SWS | 66.88 [57.78 to 75.98] | 34.78 [25.87 to 43.69] | 45.95 [36.85 to 55.06]
  Stage R Sleep | 70.40 [64.32 to 76.48] | 51.80 [45.86 to 57.75] | 75.37 [69.29 to 81.45]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; Stage N1 sleep: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p = 0.0076, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -5.67, 95% CI 2-sided [-9.80 to -1.54], Standard Error of Mean 2.09
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -10.32, 95% CI 2-sided [-14.43 to -6.21], Standard Error of Mean 2.08
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0257, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean difference = 4.65, 95% CI 2-sided [0.58 to 8.73], Standard Error of Mean 2.06
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Stage N2 sleep: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 22.70, 95% CI 2-sided [10.74 to 34.67], Standard Error of Mean 6.05
Statistical Analysis 5: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.0174, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -14.47, 95% CI 2-sided [-26.35 to -2.59], Standard Error of Mean 6.00
Statistical Analysis 6: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 37.17, 95% CI 2-sided [25.38 to 48.96], Standard Error of Mean 5.96
Statistical Analysis 7: Comparison: Pregabalin 300 mg vs Placebo; Stage N3 sleep/SWS: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 20.93, 95% CI 2-sided [12.61 to 29.25], Standard Error of Mean 4.20
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — This analysis was step 4 in a step-down procedure (if p-value < 0.05, then continue to next step) used to control the Type I error rate; LS Mean Difference = 32.10, 95% CI 2-sided [23.83 to 40.36], Standard Error of Mean 4.18
Statistical Analysis 9: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.0080, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -11.17, 95% CI 2-sided [-19.37 to -2.97], Standard Error of Mean 4.14
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; Stage R sleep: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p = 0.0834, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -4.97, 95% CI 2-sided [-10.61 to 0.67], Standard Error of Mean 2.85
Statistical Analysis 11: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 18.59, 95% CI 2-sided [12.99 to 24.19], Standard Error of Mean 2.83
Statistical Analysis 12: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -23.56, 95% CI 2-sided [-29.12 to -18.01], Standard Error of Mean 2.81

5. Secondary Outcome: Number of Awakenings of at Least 1 Epoch After Sleep Onset (NAASO1)
Description: NAASO1, as determined by PSG, was the number of times there was a wake period of at least 1 epoch from the onset of persistent sleep to light on. Each entry to be counted must be separated by a Stage 2 Non-REM [Stage N2] 30-second (30-sec) epoch, Stage 3 Non-REM [Stage N3] 30-sec epoch, or stage rapid eye movement [stage R] 30-sec epoch. The sum of 2 consecutive days of recording was divided by 2 at the end of each intervention period. Arithmetic mean of NAASO1 of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: awakenings
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
awakenings | 18.43 [16.49 to 20.36] | 26.30 [24.41 to 28.19] | 21.10 [19.16 to 23.04]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0077, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -2.67, 95% CI 2-sided [-4.63 to -0.72], Standard Error of Mean 0.99
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — This analysis was step 5 in a step-down procedure (if p-value < 0.05, then continue to next step) used to control the Type I error rate; LS Mean Difference = -7.87, 95% CI 2-sided [-9.81 to -5.93], Standard Error of Mean 0.98
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 5.20, 95% CI 2-sided [3.27 to 7.12], Standard Error of Mean 0.97

6. Secondary Outcome: Restless Legs Syndrome-Next Day Impact (RLS-NDI)
Description: RLS-NDI:participant-rated instrument to assess daytime performance and participant's previous night's sleep, consists of 14 items encompassing 5 domains:tiredness;emotional functioning;social functioning;cognitive functioning;activities of daily living and 1 global item for overall well-being. Each item: 0-10 scale; 0=Not at all; 10=Extremely. Total score: sum of scores from question 1-14 (question 10, 11: scores reversed). Total score range: 0-140; higher scores: more severe impact. Arithmetic mean of RLS-NDI of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: Week 3 and Week 5 of Each Intervention Period or ET
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 72 | 70
units on a scale | 41.43 [35.36 to 47.50] | 46.33 [40.39 to 52.27] | 46.78 [40.75 to 52.81]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0396, Mixed Models Analysis — This analysis was step 6 in a step-down procedure (if p-value < 0.05, then continue to next step) used to control the Type I error rate; LS Mean Difference = -5.35, 95% CI 2-sided [-10.44 to -0.26], Standard Error of Mean 2.57
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0568, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -4.90, 95% CI 2-sided [-9.95 to 0.14], Standard Error of Mean 2.55
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8589, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.45, 95% CI 2-sided [-5.44 to 4.54], Standard Error of Mean 2.52

7. Secondary Outcome: Periodic Limb Movement Index (PLMI)
Description: PLMI, as determined by PSG was number of periodic limb movements per hour based on time in bed (TIB). Arithmetic mean of PLMI of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: movement/hour
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
movement/hour | 25.45 [20.99 to 29.91] | 14.11 [9.79 to 18.42] | 39.95 [35.48 to 44.41]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -14.50, 95% CI 2-sided [-20.26 to -8.74], Standard Error of Mean 2.91
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 11.35, 95% CI 2-sided [5.65 to 17.04], Standard Error of Mean 2.88
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -25.84, 95% CI 2-sided [-31.51 to -20.17], Standard Error of Mean 2.86

8. Secondary Outcome: Periodic Limb Movement in Sleep Index (PLMSI)
Description: PLMSI, as determined by PSG was number of periodic limb movements in sleep per hour based on TST. Arithmetic mean of PLMSI of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: movement/hour
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
movement/hour | 22.42 [17.46 to 27.39] | 8.00 [3.20 to 12.80] | 36.95 [31.99 to 41.92]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -14.53, 95% CI 2-sided [-20.84 to -8.22], Standard Error of Mean 3.19
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 14.42, 95% CI 2-sided [8.18 to 20.67], Standard Error of Mean 3.15
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -28.95, 95% CI 2-sided [-35.16 to -22.74], Standard Error of Mean 3.14

9. Secondary Outcome: Number of Awakenings of at Least 2 Epochs After Sleep Onset (NAASO2)
Description: NAASO2, as determined by PSG, was the number of times there was a wake period of at least 2 30-sec epochs from the onset of persistent sleep to light on. Each entry to be counted must be separated by a Stage N2 30-sec epoch, Stage N3 30-sec epoch, or Stage R 30-sec epoch. The sum of 2 consecutive days of recording was divided by 2 at the end of each intervention period. Arithmetic mean of NAASO2 of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: awakenings
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
awakenings | 7.68 [6.55 to 8.82] | 12.39 [11.28 to 13.50] | 10.55 [9.42 to 11.68]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -2.86, 95% CI 2-sided [-3.93 to -1.80], Standard Error of Mean 0.54
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -4.71, 95% CI 2-sided [-5.76 to -3.65], Standard Error of Mean 0.53
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 1.84, 95% CI 2-sided [0.79 to 2.89], Standard Error of Mean 0.53

10. Secondary Outcome: Number of Arousals (NASO)
Description: NASO, as determined by PSG, was calculated as number of times there is a shift from a stage N2 to N3 or R 30-sec epoch to a stage N1 30-sec epoch from the onset of persistent sleep to light on. The sum of 2 consecutive days of recording was divided by 2 at the end of each intervention period. Arithmetic mean of NASO of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: arousals
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
arousals | 17.84 [15.06 to 20.61] | 24.19 [21.47 to 26.90] | 20.29 [17.51 to 23.06]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0617, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -2.45, 95% CI 2-sided [-5.02 to 0.12], Standard Error of Mean 1.30
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -6.35, 95% CI 2-sided [-8.91 to -3.80], Standard Error of Mean 1.29
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0028, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 3.90, 95% CI 2-sided [1.37 to 6.44], Standard Error of Mean 1.28

11. Secondary Outcome: Arousal Index (NASOI)
Description: Arousal index, as determined by PSG, was NASO per hours of sleep from the onset of persistent sleep to light on. Arithmetic mean of NASOI of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: arousals/hour
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
arousals/hour | 2.75 [2.23 to 3.28] | 4.18 [3.67 to 4.69] | 3.44 [2.92 to 3.96]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0056, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.69, 95% CI 2-sided [-1.17 to -0.21], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -1.42, 95% CI 2-sided [-1.90 to -0.95], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0026, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.74, 95% CI 2-sided [0.26 to 1.21], Standard Error of Mean 0.24

12. Secondary Outcome: International Restless Legs Syndrome Study Group Rating Scale (IRLS)
Description: IRLS: psychometrically; clinically valid; clinician-administered instrument assesses severity of RLS. RLS symptom severity and impact on daily living comprise of 10 items giving 2 subscale scores and 1 global score. Subscale scores: symptom severity(6 items) and impact on daily living(3 items), item 3 loaded equally on both subscales. Global score calculated from 10 items. Score of all items range from 0-4, total score range:0-40. Lower scores: lower severity and better quality of life. Arithmetic mean of IRLS of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 68 | 70 | 69
units on a scale | 12.28 [10.32 to 14.24] | 15.35 [13.42 to 17.28] | 18.38 [16.42 to 20.34]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -6.10, 95% CI 2-sided [-8.10 to -4.09], Standard Error of Mean 1.01
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -3.07, 95% CI 2-sided [-5.07 to -1.07], Standard Error of Mean 1.01
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0032, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -3.03, 95% CI 2-sided [-5.02 to -1.04], Standard Error of Mean 1.01

13. Secondary Outcome: Percentage of Participants With Response to Clinical Global Impression - Improvement (CGI-I) Scale
Description: CGI-I: 7-point clinician rated scale to assess improvement in disease condition as compared to the start of the study medication (baseline), ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved). Higher score = more affected.
Time Frame: Baseline, Week 5 (End of Intervention Period 1), Week 11 (End of Intervention Period 2) and Week 17 (End of Intervention Period 3) or ET
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 70 | 69
percentage of participants | 61.2 | 50.0 | 33.3

14. Secondary Outcome: Latency to Stage R Sleep (LREM)
Description: LREM, as determined by PSG, was number of non-wake epochs from the beginning of the recording to the first occurrence of Stage R sleep divided by 2. Arithmetic mean of LREM of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
minutes | 95.22 [82.11 to 108.33] | 130.99 [118.26 to 143.72] | 84.52 [71.40 to 97.64]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1677, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 10.69, 95% CI 2-sided [-4.56 to 25.95], Standard Error of Mean 7.71
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -35.77, 95% CI 2-sided [-50.88 to -20.66], Standard Error of Mean 7.63
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 46.47, 95% CI 2-sided [31.45 to 61.48], Standard Error of Mean 7.59

15. Secondary Outcome: Latency to Persistent Sleep (LPS)
Description: LPS, as determined by PSG, was number of epochs from the beginning of the recording ("lights-out") to the start of the first 20 consecutive non-wake epochs (10 minutes of persistent sleep) divided by 2. Arithmetic mean of LPS of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
minutes | 31.13 [22.06 to 40.19] | 31.52 [22.68 to 40.36] | 38.86 [29.78 to 47.93]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1040, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -7.73, 95% CI 2-sided [-17.07 to 1.61], Standard Error of Mean 4.72
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9325, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.40, 95% CI 2-sided [-9.67 to 8.87], Standard Error of Mean 4.68
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1175, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -7.33, 95% CI 2-sided [-16.54 to 1.87], Standard Error of Mean 4.65

16. Secondary Outcome: Wake Time During Sleep (WTDS)
Description: WTDS, as determined by PSG, was the number of wake (30-sec) epochs after the onset of persistent sleep and prior to the final awakening or at the end of 8-hour recording. WTDS was the sum of 2 consecutive days of recordings divided by 2 at the end of each intervention period. Arithmetic mean of WTDS of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
minutes | 45.77 [37.81 to 53.73] | 70.51 [62.77 to 78.25] | 69.75 [61.78 to 77.72]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -23.98, 95% CI 2-sided [-32.78 to -15.18], Standard Error of Mean 4.45
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -24.74, 95% CI 2-sided [-33.46 to -16.02], Standard Error of Mean 4.41
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8622, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.76, 95% CI 2-sided [-7.90 to 9.43], Standard Error of Mean 4.38

17. Secondary Outcome: Wake Time After Sleep (WTAS)
Description: WTAS, as determined by PSG, was the number of wake (30-sec) epochs after the final awakening until the end of the 8-hour recording. WTAS was the sum of 2 consecutive days of recordings divided by 2 at the end of each intervention period. Arithmetic mean of WTAS of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
minutes | 5.58 [2.15 to 9.00] | 7.86 [4.53 to 11.19] | 8.88 [5.45 to 12.30]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0800, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -3.30, 95% CI 2-sided [-7.00 to 0.40], Standard Error of Mean 1.87
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2209, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -2.28, 95% CI 2-sided [-5.95 to 1.39], Standard Error of Mean 1.86
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5815, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -1.02, 95% CI 2-sided [-4.66 to 2.63], Standard Error of Mean 1.84

18. Secondary Outcome: Total Sleep Time (TST)
Description: TST, as determined by PSG, was the number of non-wake (30-sec) epochs from the beginning of recording to the end of the recording. TST was the sum of 2 consecutive days of recording divided by 2 at the end of each intervention period. Arithmetic mean of TST of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
minutes | 402.38 [390.60 to 414.15] | 376.52 [364.99 to 388.05] | 369.66 [357.88 to 381.44]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 32.72, 95% CI 2-sided [22.02 to 43.42], Standard Error of Mean 5.41
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 25.86, 95% CI 2-sided [15.22 to 36.49], Standard Error of Mean 5.37
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2005, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 6.86, 95% CI 2-sided [-3.69 to 17.42], Standard Error of Mean 5.33

19. Secondary Outcome: Sleep Efficiency (SE)
Description: SE, as determined by PSG, was the TST divided by the time in bed (TIB)(both in minutes), multiplied by 100. Sum of 2 consecutive days of recording divided by 2 at the end of each intervention period. Arithmetic mean of SE of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of time asleep
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
Percentage of time asleep | 83.81 [81.36 to 86.27] | 78.58 [76.17 to 80.98] | 77.02 [74.56 to 79.48]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 6.80, 95% CI 2-sided [4.57 to 9.02], Standard Error of Mean 1.12
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 5.24, 95% CI 2-sided [3.02 to 7.45], Standard Error of Mean 1.12
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1622, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 1.56, 95% CI 2-sided [-0.64 to 3.75], Standard Error of Mean 1.11

20. Secondary Outcome: Hourly and Quarterly Assessment of Wake After Sleep Onset (WASO)
Description: WASO, as determined by PSG was time spent awake from sleep onset to final awakening. WASO = (sum of WTDS 30-sec epochs and WTAS 30-sec epochs)/2, measured on 2 consecutive days at end of each intervention period by each individual hour (8 hours total) and each individual quarter of night (eight hours in 2 hour increments). Arithmetic mean of WASO of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: ITT population included set of randomized participants who had at least 1 dose of study medication and had at least 1 post-randomization efficacy assessment. Here "n" signifies number of participants analyzed at that particular time point for each arm group respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 73 | 76 | 72
minutes
  Hour 1 (n= 66, 67, 66) | 1.62 (4.12) [0.70 to 2.54] | 2.26 (2.69) [1.35 to 3.17] | 3.35 (3.84) [2.41 to 4.28]
  Hour 2 (n= 67, 70, 66) | 5.04 (6.15) [3.54 to 6.53] | 7.07 (5.48) [5.61 to 8.53] | 7.39 (6.85) [5.86 to 8.93]
  Hour 3 (n= 67, 70, 67) | 4.89 [3.14 to 6.64] | 8.23 [6.52 to 9.93] | 8.90 [7.13 to 10.68]
  Hour 4 (n= 67, 70, 68) | 6.21 [4.29 to 8.13] | 11.54 [9.67 to 13.42] | 9.52 [7.59 to 11.44]
  Hour 5 (n= 67, 70, 68) | 5.93 [3.80 to 8.06] | 10.39 [8.32 to 12.46] | 10.04 [7.91 to 12.17]
  Hour 6 (n= 67, 71, 68) | 5.78 [3.49 to 8.08] | 10.54 [8.32 to 12.76] | 10.52 [8.22 to 12.81]
  Hour 7 (n= 67, 71, 68) | 9.18 [6.72 to 11.64] | 11.44 [9.06 to 13.82] | 12.09 [9.63 to 14.55]
  Hour 8 (n= 67, 71, 68) | 13.16 [10.09 to 16.23] | 18.27 [15.28 to 21.25] | 18.15 [15.08 to 21.22]
  Quarter 1 (n= 67, 70, 66) | 6.42 [4.59 to 8.26] | 8.99 [7.20 to 10.78] | 10.35 [8.47 to 12.23]
  Quarter 2 (n= 67, 70, 68) | 11.08 [8.09 to 14.07] | 19.77 [16.86 to 22.69] | 18.18 [15.19 to 21.17]
  Quarter 3 (n= 67, 71, 68) | 11.81 [8.03 to 15.59] | 20.77 [17.11 to 24.42] | 20.55 [16.77 to 24.33]
  Quarter 4 (n= 67, 71, 68) | 22.37 [17.70 to 27.04] | 29.55 [25.00 to 34.10] | 30.21 [25.54 to 34.89]

21. Secondary Outcome: Hourly and Quarterly Assessment of Number of Awakenings of at Least 1 Epoch After Sleep Onset (NAASO1)
Description: NAASO1, as determined by PSG, was the number of times there was a wake period of at least 1 30-sec epoch from the onset of persistent sleep to light on. Each entry to be counted must be separated by a Stage N2 30-sec epoch, Stage N3 30-sec epoch, or Stage R 30-sec epoch. The sum of 2 consecutive days of recording was divided by 2 at the end of each intervention period by each individual hour (8 hours total) and each individual quarter of the night (eight hours in 2 hour increments). Arithmetic mean of NAASO1 of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 20
Measure: Least Squares Mean (95% Confidence Interval); unit: awakenings
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 73 | 76 | 72
awakenings
  Hour 1 (n= 66, 67, 66) | 0.70 (0.90) [0.47 to 0.93] | 1.39 (1.12) [1.16 to 1.62] | 1.10 (0.76) [0.87 to 1.34]
  Hour 2 (n= 67, 70, 66) | 2.06 (1.41) [1.68 to 2.44] | 3.32 (1.74) [2.96 to 3.69] | 2.47 (1.44) [2.09 to 2.86]
  Hour 3 (n= 67, 70, 67) | 2.09 [1.69 to 2.48] | 3.42 [3.03 to 3.81] | 2.66 [2.25 to 3.06]
  Hour 4 (n= 67, 70, 68) | 2.44 [2.00 to 2.88] | 3.83 [3.40 to 4.25] | 2.71 [2.27 to 3.15]
  Hour 5 (n= 67, 70, 68) | 2.47 [2.06 to 2.89] | 3.76 [3.36 to 4.17] | 2.87 [2.46 to 3.29]
  Hour 6 (n= 67, 71, 68) | 2.91 [2.46 to 3.36] | 3.68 [3.24 to 4.12] | 3.16 [2.71 to 3.62]
  Hour 7 (n= 67, 71, 68) | 3.07 [2.62 to 3.53] | 4.04 [3.60 to 4.47] | 3.32 [2.87 to 3.77]
  Hour 8 (n= 67, 71, 68) | 2.76 [2.30 to 3.21] | 3.46 [3.02 to 3.90] | 3.11 [2.65 to 3.56]
  Quarter 1 (n= 67, 70, 66) | 2.71 [2.22 to 3.20] | 4.61 [4.13 to 5.09] | 3.49 [2.98 to 3.99]
  Quarter 2 (n= 67, 70, 68) | 4.53 [3.86 to 5.21] | 7.27 [6.61 to 7.93] | 5.32 [4.64 to 5.99]
  Quarter 3 (n= 67, 71, 68) | 5.39 [4.66 to 6.12] | 7.37 [6.66 to 8.08] | 6.04 [5.31 to 6.77]
  Quarter 4 (n= 67, 71, 68) | 5.87 [5.15 to 6.59] | 7.36 [6.67 to 8.06] | 6.44 [5.73 to 7.16]

22. Secondary Outcome: Hourly and Quarterly Assessment of Number of Awakenings of at Least 2 Epoch After Sleep Onset (NAASO2)
Description: NAASO2, as determined by PSG, was the number of times there was a wake period of at least 2 30-sec epochs from the onset of persistent sleep to light on. Each entry to be counted must be separated by a Stage N2 30-sec epoch, Stage N3 30-sec epoch, or Stage R 30-sec epoch. The sum of 2 consecutive days of recording was divided by 2 at the end of each intervention period by each individual hour (8 hours total) and each individual quarter of the night (eight hours in 2 hour increments). Arithmetic mean of NAASO2 of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 20
Measure: Least Squares Mean (95% Confidence Interval); unit: awakenings
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 73 | 76 | 72
awakenings
  Hour 1 (n= 66, 67, 66) | 0.42 (0.60) [0.26 to 0.58] | 0.61 (0.71) [0.45 to 0.76] | 0.73 (0.59) [0.57 to 0.89]
  Hour 2 (n= 67, 70, 66) | 1.04 (0.83) [0.79 to 1.29] | 1.72 (1.13) [1.48 to 1.96] | 1.37 (1.06) [1.12 to 1.63]
  Hour 3 (n= 67, 70, 67) | 0.99 [0.75 to 1.23] | 1.71 [1.48 to 1.95] | 1.41 [1.17 to 1.65]
  Hour 4 (n= 67, 70, 68) | 1.01 [0.74 to 1.27] | 1.84 [1.58 to 2.09] | 1.48 [1.22 to 1.74]
  Hour 5 (n= 67, 70, 68) | 1.06 [0.81 to 1.31] | 1.76 [1.52 to 2.01] | 1.48 [1.22 to 1.73]
  Hour 6 (n= 67, 71, 68) | 1.02 [0.79 to 1.26] | 1.57 [1.34 to 1.80] | 1.44 [1.20 to 1.68]
  Hour 7 (n= 67, 71, 68) | 1.24 [0.97 to 1.51] | 1.94 [1.68 to 2.20] | 1.57 [1.30 to 1.84]
  Hour 8 (n= 67, 71, 68) | 1.00 [0.75 to 1.24] | 1.56 [1.32 to 1.79] | 1.28 [1.04 to 1.52]
  Quarter 1 (n= 67, 70, 66) | 1.43 [1.11 to 1.75] | 2.27 [1.96 to 2.58] | 2.06 [1.73 to 2.38]
  Quarter 2 (n= 67, 70, 68) | 1.99 [1.58 to 2.39] | 3.56 [3.16 to 3.96] | 2.85 [2.44 to 3.26]
  Quarter 3 (n= 67, 71, 68) | 2.10 [1.68 to 2.51] | 3.30 [2.89 to 3.70] | 2.92 [2.50 to 3.34]
  Quarter 4 (n= 67, 71, 68) | 2.25 [1.86 to 2.64] | 3.44 [3.06 to 3.82] | 2.86 [2.47 to 3.25]

23. Secondary Outcome: Hourly and Quarterly Assessment of Number of Arousals (NASO)
Description: NASO, as determined by PSG was the number of times there is a shift from a stage N2 to N3 or R 30-sec epoch to a stage N1 30-sec epoch from the onset of persistent sleep to light on. The sum of 2 consecutive days of recording was divided by 2 at the end of each intervention period by each individual hour (8 hours total) and each individual quarter of the night (eight hours in 2 hour increments). Arithmetic mean of NASO for each participant at each period was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 20
Measure: Least Squares Mean (95% Confidence Interval); unit: arousals
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 73 | 76 | 72
arousals
  Hour 1 (n= 66, 67, 66) | 1.48 (1.65) [1.01 to 1.94] | 2.06 (2.22) [1.60 to 2.52] | 1.79 (1.78) [1.32 to 2.26]
  Hour 2 (n= 67, 70, 66) | 2.36 (2.03) [1.85 to 2.86] | 3.23 (2.15) [2.74 to 3.72] | 2.68 (1.99) [2.16 to 3.19]
  Hour 3 (n= 67, 70, 67) | 2.31 [1.75 to 2.87] | 3.23 [2.68 to 3.78] | 2.80 [2.23 to 3.37]
  Hour 4 (n= 67, 70, 68) | 2.94 [2.39 to 3.49] | 3.41 [2.88 to 3.94] | 2.76 [2.22 to 3.31]
  Hour 5 (n= 67, 70, 68) | 2.33 [1.76 to 2.90] | 3.20 [2.64 to 3.75] | 2.89 [2.32 to 3.46]
  Hour 6 (n= 67, 71, 68) | 2.39 [1.88 to 2.90] | 3.30 [2.80 to 3.80] | 2.70 [2.19 to 3.22]
  Hour 7 (n= 67, 71, 68) | 2.15 [1.67 to 2.63] | 3.28 [2.81 to 3.75] | 2.66 [2.18 to 3.14]
  Hour 8 (n= 67, 71, 68) | 2.07 [1.56 to 2.57] | 2.98 [2.49 to 3.46] | 2.46 [1.96 to 2.97]
  Quarter 1 (n= 67, 70, 66) | 3.75 [2.93 to 4.57] | 5.09 [4.28 to 5.89] | 4.26 [3.43 to 5.09]
  Quarter 2 (n= 67, 70, 68) | 5.25 [4.32 to 6.18] | 6.67 [5.76 to 7.57] | 5.55 [4.62 to 6.48]
  Quarter 3 (n= 67, 71, 68) | 4.75 [3.86 to 5.64] | 6.44 [5.58 to 7.30] | 5.61 [4.72 to 6.50]
  Quarter 4 (n= 67, 71, 68) | 4.23 [3.39 to 5.06] | 6.24 [5.43 to 7.04] | 5.13 [4.29 to 5.96]

24. Secondary Outcome: Hourly and Quarterly Assessment of Periodic Limb Movement (PLM)
Description: PLM, as determined by PSG was number of periodic limb movements based on time in bed (TIB). Calculated at each individual hour (8 hours total) and each individual quarter of the night (eight hours in 2 hour increments). Arithmetic mean of PLM of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: ITT population included set of randomized participants who had at least one dose of study medication and had at least one post-randomization efficacy assessment. 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: movement/hour
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
movement/hour
  Hour 1 | 31.45 (29.70) [23.60 to 39.30] | 21.57 (27.03) [13.96 to 29.18] | 54.67 (39.98) [46.81 to 62.53]
  Hour 2 | 26.38 (29.20) [19.25 to 33.51] | 12.49 (14.51) [5.59 to 19.39] | 52.93 (40.92) [45.80 to 60.07]
  Hour 3 | 40.93 [32.38 to 49.48] | 14.05 [5.77 to 22.32] | 48.76 [40.20 to 57.32]
  Hour 4 | 30.35 [23.05 to 37.64] | 14.50 [7.45 to 21.55] | 46.58 [39.29 to 53.88]
  Hour 5 | 25.70 [19.02 to 32.38] | 11.93 [5.47 to 18.38] | 36.17 [29.49 to 42.86]
  Hour 6 | 21.02 [15.01 to 27.04] | 10.57 [4.75 to 16.38] | 32.47 [26.45 to 38.49]
  Hour 7 | 14.22 [9.06 to 19.37] | 11.11 [6.12 to 16.09] | 27.04 [21.88 to 32.20]
  Hour 8 | 13.37 [8.54 to 18.20] | 16.55 [11.86 to 21.24] | 20.97 [16.14 to 25.81]
  Quarter 1 | 57.82 [44.51 to 71.12] | 34.02 [21.14 to 46.91] | 107.56 [94.24 to 120.87]
  Quarter 2 | 71.29 [56.94 to 85.64] | 28.55 [14.66 to 42.43] | 95.31 [80.95 to 109.67]
  Quarter 3 | 46.77 [35.42 to 58.11] | 22.49 [11.51 to 33.46] | 68.66 [57.30 to 80.01]
  Quarter 4 | 27.60 [18.97 to 36.24] | 27.64 [19.28 to 36.00] | 48.01 [39.36 to 56.65]

25. Secondary Outcome: Hourly and Quarterly Assessment of Sleep Efficiency (SE)
Description: SE, as determined by PSG, was the TST divided by the time in bed (TIB)(both in minutes), multiplied by 100. Sum of 2 consecutive days of recording divided by 2 at the end of each intervention period by each individual hour (8 hours total) and each individual quarter of the night (eight hours in 2 hour increments). Arithmetic mean for SE of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 24
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of time asleep
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 71 | 68
percentage of time asleep
  Hour 1 | 62.31 (24.14) [56.62 to 68.01] | 66.88 (24.30) [61.33 to 72.43] | 57.80 (22.90) [52.10 to 63.49]
  Hour 2 | 86.13 (16.94) [81.85 to 90.41] | 83.43 (16.03) [79.26 to 87.60] | 77.31 (20.49) [73.03 to 81.60]
  Hour 3 | 90.22 [86.68 to 93.77] | 84.86 [81.43 to 88.29] | 81.86 [78.32 to 85.40]
  Hour 4 | 89.41 [85.86 to 92.97] | 79.84 [76.40 to 83.28] | 82.61 [79.05 to 86.16]
  Hour 5 | 90.00 [86.30 to 93.70] | 81.85 [78.27 to 85.43] | 82.92 [79.22 to 86.63]
  Hour 6 | 90.33 [86.45 to 94.21] | 81.64 [77.88 to 85.39] | 82.49 [78.61 to 86.38]
  Hour 7 | 84.70 [80.60 to 88.80] | 80.90 [76.92 to 84.87] | 79.86 [75.76 to 83.96]
  Hour 8 | 78.07 [72.95 to 83.19] | 69.51 [64.53 to 74.50] | 69.75 [64.63 to 74.88]
  Quarter 1 | 74.21 [69.69 to 78.73] | 75.15 [70.73 to 79.57] | 67.62 [63.10 to 72.15]
  Quarter 2 | 89.84 [86.77 to 92.92] | 82.37 [79.38 to 85.35] | 82.30 [79.23 to 85.38]
  Quarter 3 | 90.09 [86.83 to 93.34] | 81.74 [78.59 to 84.90] | 82.75 [79.49 to 86.01]
  Quarter 4 | 81.37 [77.45 to 85.28] | 75.16 [71.35 to 78.97] | 74.84 [70.93 to 78.76]

26. Secondary Outcome: Subjective Sleep Questionnaire (SSQ): Number of Awakenings Subscale
Description: SSQ: participant-rated instrument to assess sleep behavior; measures sleep quantity, quality. Comprised of 5 items giving 5 subscale scores: latency, hours of sleep, number of awakenings, total wake time after sleep onset, quality of sleep. This (1 item) subscale: numerical rating completed by participant 30 minutes after waking; recall period: night before. Range: 0 awakenings to 30 awakenings. Lower value indicates better quality of sleep. Arithmetic mean of this subscale score of each participant for all periods was taken prior to employing linear mixed model. Results of hours of sleep subscale reported as sTST.
Time Frame: Week 3 and Week 5 of Each Intervention Period or ET
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: awakenings
Groups:
- Placebo: PBO capsule matched to PPX 0.5 mg once daily in any intervention period.
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 72 | 70
awakenings | 1.69 [1.34 to 2.03] | 2.64 [2.31 to 2.98] | 2.51 [2.17 to 2.86]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.83, 95% CI 2-sided [-1.18 to -0.47], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.96, 95% CI 2-sided [-1.31 to -0.60], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.4677, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.13, 95% CI 2-sided [-0.22 to 0.48], Standard Error of Mean 0.18

27. Secondary Outcome: Subjective Sleep Questionnaire (SSQ): Total Wake Time After Sleep Onset Subscale
Description: SSQ: participant-rated instrument to assess sleep behavior; measures sleep quantity, quality. Comprised of 5 items yielding 5 subscale scores: latency, hours of sleep, number of awakenings, total wake time after sleep onset, quality of sleep. This 1 item subscale (in minutes): numerical rating completed by participant 30 minutes after waking; recall period: night before. Range: 0-1440 minutes. Lower value: better sleep. Arithmetic mean of this subscale score of each participant for all periods was taken prior to employing linear mixed model. Results of hours of sleep subscale reported as sTST.
Time Frame: Week 3 and Week 5 of each intervention period or ET
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 65 | 71 | 70
minutes | 53.78 [42.94 to 64.61] | 82.23 [71.76 to 92.70] | 79.09 [68.46 to 89.72]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -25.32, 95% CI 2-sided [-35.83 to -14.80], Standard Error of Mean 5.31
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -28.45, 95% CI 2-sided [-38.89 to -18.02], Standard Error of Mean 5.27
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5461, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 3.14, 95% CI 2-sided [-7.13 to 13.40], Standard Error of Mean 5.19

28. Secondary Outcome: Subjective Sleep Questionnaire (SSQ): Quality of Sleep Subscale
Description: SSQ: participant-rated instrument to assess sleep behavior; measures sleep quantity, quality. Comprised of 5 items yielding 5 subscale scores: latency, hours of sleep, number of awakenings, total wake time after sleep onset, quality of sleep. This 1 item subscale: numerical rating completed by participant 30 minutes after waking; recall period: night before, Range: 0 to 100, higher score: better quality of sleep. Arithmetic mean of this subscale score of each participant for all periods was taken prior to employing linear mixed model. Results of hours of sleep subscale reported as sTST.
Time Frame: Week 3 and Week 5 of each intervention period or ET
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 72 | 70
units on a scale | 6.74 [6.35 to 7.13] | 5.69 [5.31 to 6.06] | 5.70 [5.32 to 6.08]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 1.04, 95% CI 2-sided [0.63 to 1.45], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 1.05, 95% CI 2-sided [0.65 to 1.46], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9403, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.02, 95% CI 2-sided [-0.42 to 0.39], Standard Error of Mean 0.20

29. Secondary Outcome: Subjective Sleep Questionnaire (SSQ): Latency Subscale
Description: SSQ: participant-rated instrument assesses sleep behavior; measures sleep quantity, quality. Comprised of 5 items giving 5 subscale scores: latency, hours of sleep, number of awakenings, total wake time after sleep onset, quality of sleep. Latency (time to fall asleep [in minutes]): numerical rating completed by participant 30 minutes after waking; recall period: night before. Range: 0 - 840 minutes, lower value: better sleep. Arithmetic mean of subscale score of each participant for all periods was taken prior to employing linear mixed model. Hours of sleep subscale results reported as sTST.
Time Frame: Week 3 and Week 5 of each intervention period or ET
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 67 | 72 | 70
minutes | 42.49 [34.26 to 50.72] | 40.59 [32.52 to 48.66] | 50.07 [41.89 to 58.25]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0215, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -7.58, 95% CI 2-sided [-14.03 to -1.14], Standard Error of Mean 3.26
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5569, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 1.90, 95% CI 2-sided [-4.49 to 8.29], Standard Error of Mean 3.23
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0036, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -9.48, 95% CI 2-sided [-15.81 to -3.16], Standard Error of Mean 3.20

30. Secondary Outcome: Medical Outcomes Study - Sleep Scale (MOS-SS)
Description: MOS-SS:Participant rated instrument, assesses sleep quantity, quality;with 12 items(7 subscale scores:sleep disturbance, snoring, awakening short of breath/with headache, sleep adequacy, somnolence, sleep quantity, optimal sleep;2 composite index scores:sleep problems Index I, II). Subscale scores total range:0-100(except sleep quantity[range 0-24 hours], optimal sleep[range 0-1: 0= <7 or >8 hours;1=7/8 hours]). Higher scores=poorer sleep outcomes(except sleep quantity, adequacy). Arithmetic mean of MOS-SS scores of each participant for all periods was taken before linear mixed model analysis.
Time Frame: as for outcome 2
Population: ITT population included set of randomized participants who had at least 1 dose of study medication and had at least 1 post-randomization efficacy assessment. Here "n" signifies number of participants analyzed for particular subscale for each arm group respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 73 | 76 | 72
units on a scale
  Awaken Short of Breath/with Headache (n= 68,71,69) | 11.59 [6.20 to 16.97] | 13.10 [7.77 to 18.44] | 10.88 [5.49 to 16.27]
  Adequacy (n= 68,71,69) | 54.96 [48.11 to 61.81] | 43.90 [37.21 to 50.58] | 40.79 [33.93 to 47.65]
  Somnolence (n= 68,71,69) | 21.28 [17.08 to 25.47] | 21.32 [17.21 to 25.44] | 23.71 [19.51 to 27.90]
  Sleep Quantity (n= 68,71,69) | 6.43 [5.95 to 6.91] | 6.50 [6.03 to 6.97] | 5.97 [5.49 to 6.46]
  6-Item Sleep Problems Index (n= 68,71,69) | 30.69 [25.94 to 35.45] | 37.24 [32.58 to 41.89] | 40.59 [35.83 to 45.34]
  9-Item Sleep Problems Index (n= 68,71,69) | 32.75 [28.06 to 37.44] | 37.88 [33.28 to 42.47] | 42.89 [38.20 to 47.59]
  Optimal Sleep (n= 68,71,69) | 0.43 [0.32 to 0.54] | 0.35 [0.24 to 0.46] | 0.29 [0.18 to 0.40]
  Sleep Disturbance (n= 68,71,69) | 34.08 [28.11 to 40.06] | 40.19 [34.34 to 46.04] | 48.65 [42.66 to 54.63]
  Snoring (n= 67,71,68) | 15.27 [10.05 to 20.49] | 15.97 [10.86 to 21.08] | 17.96 [12.75 to 23.17]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; Awaken Short of Breath/with Headache: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p = 0.6947, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.71, 95% CI 2-sided [-2.85 to 4.27], Standard Error of Mean 1.80
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 30, analysis 1]; Test type: Superiority or Other; p = 0.3980, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -1.52, 95% CI 2-sided [-5.06 to 2.02], Standard Error of Mean 1.79
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 30, analysis 1]; Test type: Superiority or Other; p = 0.2144, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 2.23, 95% CI 2-sided [-1.30 to 5.76], Standard Error of Mean 1.78
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Adequacy: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 14.17, 95% CI 2-sided [6.25 to 22.08], Standard Error of Mean 4.00
Statistical Analysis 5: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 30, analysis 4]; Test type: Superiority or Other; p = 0.0061, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 11.07, 95% CI 2-sided [3.22 to 18.92], Standard Error of Mean 3.97
Statistical Analysis 6: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 30, analysis 4]; Test type: Superiority or Other; p = 0.4342, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 3.10, 95% CI 2-sided [-4.72 to 10.93], Standard Error of Mean 3.95
Statistical Analysis 7: Comparison: Pregabalin 300 mg vs Placebo; Somnolence: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p = 0.2420, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -2.43, 95% CI 2-sided [-6.53 to 1.66], Standard Error of Mean 2.07
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 30, analysis 7]; Test type: Superiority or Other; p = 0.9810, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.05, 95% CI 2-sided [-4.12 to 4.02], Standard Error of Mean 2.05
Statistical Analysis 9: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 30, analysis 7]; Test type: Superiority or Other; p = 0.2468, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -2.38, 95% CI 2-sided [-6.44 to 1.67], Standard Error of Mean 2.05
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; Sleep Quantity: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p = 0.1496, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.46, 95% CI 2-sided [-0.17 to 1.09], Standard Error of Mean 0.32
Statistical Analysis 11: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 30, analysis 10]; Test type: Superiority or Other; p = 0.8184, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.07, 95% CI 2-sided [-0.69 to 0.55], Standard Error of Mean 0.31
Statistical Analysis 12: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 30, analysis 10]; Test type: Superiority or Other; p = 0.0918, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.53, 95% CI 2-sided [-0.09 to 1.15], Standard Error of Mean 0.31
Statistical Analysis 13: Comparison: Pregabalin 300 mg vs Placebo; 6-Item Sleep Problems Index: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -9.89, 95% CI 2-sided [-14.80 to -4.99], Standard Error of Mean 2.48
Statistical Analysis 14: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 30, analysis 13]; Test type: Superiority or Other; p = 0.0089, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -6.54, 95% CI 2-sided [-11.42 to -1.67], Standard Error of Mean 2.46
Statistical Analysis 15: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 30, analysis 13]; Test type: Superiority or Other; p = 0.1746, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -3.35, 95% CI 2-sided [-8.21 to 1.51], Standard Error of Mean 2.45
Statistical Analysis 16: Comparison: Pregabalin 300 mg vs Placebo; 9-Item Sleep Problems Index: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -10.14, 95% CI 2-sided [-14.96 to -5.32], Standard Error of Mean 2.44
Statistical Analysis 17: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 30, analysis 16]; Test type: Superiority or Other; p = 0.0359, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -5.13, 95% CI 2-sided [-9.91 to -0.34], Standard Error of Mean 2.42
Statistical Analysis 18: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 30, analysis 16]; Test type: Superiority or Other; p = 0.0395, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -5.01, 95% CI 2-sided [-9.78 to -0.24], Standard Error of Mean 2.41
Statistical Analysis 19: Comparison: Pregabalin 300 mg vs Placebo; Optimal Sleep: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p = 0.0278, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.14, 95% CI 2-sided [0.02 to 0.27], Standard Error of Mean 0.06
Statistical Analysis 20: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 30, analysis 19]; Test type: Superiority or Other; p = 0.2000, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.08, 95% CI [-0.04 to 0.20], Standard Error of Mean 0.06
Statistical Analysis 21: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 30, analysis 19]; Test type: Superiority or Other; p = 0.3396, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.06, 95% CI 2-sided [-0.06 to 0.18], Standard Error of Mean 0.06
Statistical Analysis 22: Comparison: Pregabalin 300 mg vs Placebo; Sleep Disturbance: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -14.56, 95% CI 2-sided [-20.93 to -8.19], Standard Error of Mean 3.22
Statistical Analysis 23: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 30, analysis 22]; Test type: Superiority or Other; p = 0.0584, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -6.11, 95% CI 2-sided [-12.43 to 0.22], Standard Error of Mean 3.20
Statistical Analysis 24: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 30, analysis 22]; Test type: Superiority or Other; p = 0.0090, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -8.45, 95% CI 2-sided [-14.76 to -2.15], Standard Error of Mean 3.19
Statistical Analysis 25: Comparison: Pregabalin 300 mg vs Placebo; Snoring: P-value was calculated using linear mixed model analysis with treatment, period and sequence as fixed effects. Random effects were participant within sequence and residual error. The LS means and SE were used to test for a treatment difference and construct 2-sided 95% CIs. The hypothesis test was 2-sided and conducted at the 5% level of significance; Test type: Superiority or Other; p = 0.2405, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -2.69, 95% CI 2-sided [-7.20 to 1.82], Standard Error of Mean 2.28
Statistical Analysis 26: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 30, analysis 25]; Test type: Superiority or Other; p = 0.7565, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.70, 95% CI 2-sided [-5.18 to 3.77], Standard Error of Mean 2.26
Statistical Analysis 27: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 30, analysis 25]; Test type: Superiority or Other; p = 0.3792, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -1.98, 95% CI 2-sided [-6.43 to 2.47], Standard Error of Mean 2.25

31. Secondary Outcome: Restless Leg Syndrome - Quality of Life Scale (RLS-QoL)
Description: RLS-QoL: psychometrically and clinically valid and reliable participant-rated instrument, assesses impact of RLS on participant quality of life. Specifically, it assessed effects of RLS on health status function (symptom severity, daily activity, social functioning, sleep, concentrating and decision making, travelling, sexual activity, and work) giving a summary score ranging from 0-100. Higher scores reflect better quality of life. Recall period: 1 week prior to assessment. Arithmetic mean of RLS-QoL score of each participant for all periods was taken prior to employing linear mixed model.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 68 | 71 | 69
units on a scale | 73.30 [69.72 to 76.87] | 70.05 [66.53 to 73.56] | 68.03 [64.45 to 71.61]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 5.27, 95% CI 2-sided [1.98 to 8.55], Standard Error of Mean 1.66
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0506, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 3.25, 95% CI 2-sided [-0.01 to 6.51], Standard Error of Mean 1.65
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2222, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 2.01, 95% CI 2-sided [-1.24 to 5.26], Standard Error of Mean 1.64

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. But, distinct events are presented. An event may be categorized as serious in 1 subject; as nonserious in another subject or 1 subject may have experienced both serious, nonserious events in study. 'At risk population'= who received study treatments in different interventions; PGB=75,PPX=76,PBO=73.
Groups:
- Placebo: PBO capsule matched to PPX 0.5 mg once daily or PGB 300 mg once daily (matching placebo escalation and tapering scheme was followed) in any of the intervention period.
Arm/Group | Pregabalin 300 mg | Pramipexole 0.5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/75 | 1/76 | 3/73
Other Adverse Events (participants affected / at risk) | 46/75 | 40/76 | 27/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 300 mg (N=75) | Pramipexole 0.5 mg (N=76) | Placebo (N=73)
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Blood pressure orthostatic decreased (Investigations) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 300 mg (N=75) | Pramipexole 0.5 mg (N=76) | Placebo (N=73)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Excessive eye blinking (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 4 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 6 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 1
Feeling abnormal (General disorders) | 1 | 1 | 0
Feeling drunk (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 2 | 0 | 0
Hangover (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Irritability (General disorders) | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 3 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Sinusitis (Infections and infestations) | 1 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 1 | 1
Blood pressure abnormal (Investigations) | 1 | 1 | 0
Red cell distribution width increased (Investigations) | 0 | 1 | 1
Serum ferritin decreased (Investigations) | 1 | 1 | 2
Weight increased (Investigations) | 3 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Amnesia (Nervous system disorders) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 3 | 0 | 0
Disturbance in attention (Nervous system disorders) | 4 | 0 | 0
Dizziness (Nervous system disorders) | 18 | 2 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 6 | 5
Lethargy (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 1 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0 | 0
Sedation (Nervous system disorders) | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 13 | 6 | 3
Syncope (Nervous system disorders) | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 2 | 2 | 1
Agitation (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Daydreaming (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Distractibility (Psychiatric disorders) | 1 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 0 | 1
Euphoric mood (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 2
Libido increased (Psychiatric disorders) | 0 | 1 | 0
Middle insomnia (Psychiatric disorders) | 0 | 1 | 0
Orgasm abnormal (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Renal pain (Renal and urinary disorders) | 1 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 2 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Endodontic procedure (Surgical and medical procedures) | 1 | 0 | 0
Sinus operation (Surgical and medical procedures) | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.